CLINICAL TRIAL: NCT02909140
Title: Optimal Method for Mydriasis in Cataract Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient patient recruitment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00091874
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topical Mydriasis (Experimental): Topical mydriasis will be with 1 drop of phenylephrine 2.5% and 1 drop of cyclopentolate 1% x 4 doses each, with each drop spaced 5 minutes apart given in the pre-op area. These are the standard dilating drops used for cataract surgery. These patients will also receive intracameral lidocaine 1% for anesthesia.
  Interventions: Drug: Topical phenylephrine 2.5%; Drug: Topical cyclopentolate 1%; Drug: Intracameral Lidocaine 1%
- Intracameral Mydriasis (Experimental): Intracameral mydriasis will be with 0.2ml to 0.3ml of epinephrine 1:10,000 injected into the anterior chamber at the beginning of the cataract surgery procedure. This is the standard concentration use for intracameral mydriasis in cataract surgery. These patients will also receive intracameral lidocaine 1% for anesthesia.
  Interventions: Drug: Intracameral Lidocaine 1%; Drug: Intracameral 0.2- 0.3ml of epinephrine 1:10,000
- Topical + Intracameral mydriasis (Experimental): Topical mydriasis will be with 1 drop of phenylephrine 2.5% and 1 drop of cyclopentolate 1% x 4 doses each, with each drop spaced 5 minutes apart given in the pre-op area. These are the standard dilating drops used for cataract surgery. These patients will also receive intracameral lidocaine 1% for anesthesia. Intracameral mydriasis will be with 0.2ml to 0.3ml of epinephrine 1:10,000 injected into the anterior chamber at the beginning of the cataract surgery procedure. This is the standard concentration use for intracameral mydriasis in cataract surgery. These patients will also receive intracameral lidocaine 1% for anesthesia.
  Interventions: Drug: Topical phenylephrine 2.5%; Drug: Topical cyclopentolate 1%; Drug: Intracameral Lidocaine 1%; Drug: Intracameral 0.2- 0.3ml of epinephrine 1:10,000

INTERVENTIONS:
Drug: Topical phenylephrine 2.5%
  Arms: Topical + Intracameral mydriasis; Topical Mydriasis
Drug: Topical cyclopentolate 1%
  Arms: Topical + Intracameral mydriasis; Topical Mydriasis
Drug: Intracameral Lidocaine 1%
Drug: Intracameral 0.2- 0.3ml of epinephrine 1:10,000
  Arms: Intracameral Mydriasis; Topical + Intracameral mydriasis

SUMMARY:
Obtaining appropriate mydriasis prior to cataract surgery is an important variable in successful surgery. The current practice includes using topical anticholinergic and sympathomimetic agents in the preoperative area prior to cataract surgery, but the pupils are sometimes insufficiently dilated and can often need additional mydriasis with intracameral agents during cataract surgery. Pre-operative topical mydriatic drops take time to take effect, are mildly uncomfortable for the patient, and have a cost to the healthcare system. If intracameral mydriasis alone can achieve adequate pupil dilation, perhaps topical mydriatics would not be needed. The purpose of this study is to evaluate whether topical versus intracameral versus topical + intracameral mydriasis is the optimal way to dilate pupils during routine cataract surgery. The results of this study have implications for improving the efficiency and reducing time prior to cataract surgery. In addition, it has significant potential to reduce the cost associated with cataract surgery if preoperative drops can be eliminated.

DETAILED DESCRIPTION:
Recent research has compared the use of intracameral and topical agents with the preoperative pupil size and cataract surgery success. Studies have compared topical mydriatics with intracameral lidocaine and found no significant difference in dilation. , Other studies have compared topical mydriatics with intracameral dilation that includes solutions with and without epinephrine in the irrigating solution and concluded that irrigating solutions without epinephrine can safely be used with intracameral mydriatics but epinephrine is useful when using topical mydriatics. There have also been studies comparing the success of longer acting drug inserts of mydriatic agents with the use of intracameral agents. In addition to these standard agents, different surgeons have used various formulations of topical and intracameral agents to perform mydriasis. As of yet, there is no formal, standardized method for mydriasis and no large prospective study comparing the outcomes of the various methods. Considerations such as cost and time spent on preoperative mydriatic agents in light of the amount of success seen with these agents calls into question the need for such agents. The investigators would like to study the amount of pupillary dilation seen with topical preoperative mydriatic agents compared to intracameral agents compared to the use of them both together.

This will be a prospective randomized controlled trial. Patients will be consented and enrolled at their pre-op visit. They will be randomized to topical drops alone, intracameral injection alone, or topical plus intracameral mydriasis. All patients will receive intracameral lidocaine, as this is used for its anesthetic effect but also has some mydriatic effect. The intervention will take place on the day of the operation. Patients will be followed until post-operative month #1.

Data will be gathered on 4 visits: pre-op clinic visit, day of operation, and post-operative day #1 and post-operative month #1. These are all standard visits for routine cataract surgery, and this study will not require the patient to make any extra visits. Enrollment will continue until the sample size is met.

Patients cannot be blinded to whether or not they receive topical mydriasis eyedrops, and no placebo drops are necessary because patients cannot voluntarily control their pupillary constriction, so no placebo effect would be expected. The surgeon cannot be blinded to whether or not the patient has received topical mydriasis eyedrops in the pre-op area because it will be evident based upon whether or not the patient's eye is dilated. Another researcher who was not present in the operating room will grade the photographs and measure the pupil size, and this researcher will be blinded to which intervention the patient received.

Currently, some surgeons use topical plus intracameral mydriasis for mydriasis during cataract surgery. It is hypothesized that intracameral mydriasis alone may be sufficient to adequately dilate the pupil for cataract surgery. Patients who are not adequately dilated at the time of pupil size measurement immediately before the capsulorrhexis step will subsequently receive additional pharmacologic mydriasis, visco-dilation, or iris expansion devices to dilate their pupil to a size that is adequate for their surgery. Therefore, no matter which group the patient is in, their pupil will be eventually dilated to a size that is adequate to proceed with surgery.

There is no placebo or non-treatment group, since all patients must be somehow dilated in order to undergo cataract surgery. The purpose of this study is to compare 3 methods of dilation.

The pupil size will be measured after the viscoelastic is injected and before the capsulorrhexis is performed. Treatment failure is defined as a pupil size that is clinically deemed too small to safely proceed with surgery (approximately less than 5 mm). At this point, a rescue intervention will be implemented with additional pharmacologic mydriasis, visco-dilation, or iris expansion devices, until the pupil is adequately dilated to proceed with surgery. These patients will still be included in the study, and their pupil size prior to the rescue intervention is still the primary outcome.

Participants can choose to stop participating in the study prior to receiving any of the mydriasis agents. Should they choose to withdraw from the study, they would end up receiving routine mydriasis with topical plus intracameral agents. The study ends on post-op month #1 for all individual patients. The study enrollment period will end when the sample size is met.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 40 or older who are undergoing routine cataract surgery under topical anesthesia with monitored anesthesia care at the Wilmer Eye Institute with Dr. Fasika Woreta and her senior resident proficient at cataract surgery.

Exclusion Criteria:

* Need for general anesthesia
* Maximum pupillary dilation <6.0mm at the pre-op clinic visit.
* Prior intra-ocular surgery
* Prior trauma
* Any pre-existing iris abnormalities including pupillary deformity, posterior synechiae, peripheral anterior synechiae, zonular dehiscence
* Pseudoexfoliation
* Allergy to any of the mydriasis agents
* Pregnancy or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fasika Woreta, M.D., M.P.H, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 3 patients were enrolled, no information is available for the 3rd patient. Hence, the discrepancy.
Groups:
- Topical Mydriasis: Topical mydriasis will be with 1 drop of phenylephrine 2.5% and 1 drop of cyclopentolate 1% x 4 doses each, with each drop spaced 5 minutes apart given in the pre-op area. These are the standard dilating drops used for cataract surgery. These patients will also receive intracameral lidocaine 1% for anesthesia.
  Topical phenylephrine 2.5%
  Topical cyclopentolate 1%
  Intracameral Lidocaine 1%
- Intracameral Mydriasis: Intracameral mydriasis will be with 0.2ml to 0.3ml of epinephrine 1:10,000 injected into the anterior chamber at the beginning of the cataract surgery procedure. This is the standard concentration use for intracameral mydriasis in cataract surgery. These patients will also receive intracameral lidocaine 1% for anesthesia.
  Intracameral Lidocaine 1%
  Intracameral 0.2- 0.3ml of epinephrine 1:10,000
- Topical + Intracameral Mydriasis: Topical mydriasis will be with 1 drop of phenylephrine 2.5% and 1 drop of cyclopentolate 1% x 4 doses each, with each drop spaced 5 minutes apart given in the pre-op area. These are the standard dilating drops used for cataract surgery. These patients will also receive intracameral lidocaine 1% for anesthesia. Intracameral mydriasis will be with 0.2ml to 0.3ml of epinephrine 1:10,000 injected into the anterior chamber at the beginning of the cataract surgery procedure. This is the standard concentration use for intracameral mydriasis in cataract surgery. These patients will also receive intracameral lidocaine 1% for anesthesia.
  Topical phenylephrine 2.5%
  Topical cyclopentolate 1%
  Intracameral Lidocaine 1%
  Intracameral 0.2- 0.3ml of epinephrine 1:10,000
Period: Overall Study
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Started | 0 | 2 | 0
Completed | 0 | 2 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Absent enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis | Total
Number analyzed (Participants) | 0 | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 |  | 0
  Between 18 and 65 years |  | 0 |  | 0
  >=65 years |  | 2 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 |  | 1
  Male |  | 1 |  | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Systolic blood pressure in preoperative area [Mean (Full Range); unit: mmHg] |  | 144 [140 to 148] |  | 144 [140 to 148]
Heart rate in preoperative area [Mean (Full Range); unit: bpm] |  | 75.5 [62 to 89] |  | 75.5 [62 to 89]
Systolic blood pressure on entry to OR [Mean (Full Range); unit: mmHg] |  | 172 [169 to 176] |  | 172 [169 to 176]
Heart rate on entry to OR [Mean (Full Range); unit: bpm] |  | 80.5 [72 to 89] |  | 80.5 [72 to 89]

OUTCOME MEASURES:

1. Primary Outcome: Pupil Size Immediately Prior to Capsulorrhexis
Description: Pupil size immediately prior to the capsulorrhexis step of cataract surgery. This will be recorded by digital photography and measured by a researcher who is masked to the intervention.
Time Frame: Immediately prior to the capsulorrhexis step of cataract surgery
Population: Data was only collected for the "Intracameral Mydriasis' arm. We analyzed data for 1 participant only because of lack of data for the other participant.
Measure: Number; unit: mm
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 1 | 0
mm |  | 8 |

2. Secondary Outcome: Pupil Size (mm) Immediately After Nuclear Disassembly
Description: Pupil size immediately after breaking up of cataractous lens
Time Frame: Immediately after nuclear disassembly step of cataract surgery
Population: as for outcome 1
Measure: Number; unit: mm
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 1 | 0
mm |  | 8 |

3. Secondary Outcome: Pupil Size Immediately Prior to Intraocular Lens (IOL) Insertion
Description: Pupil size after insertion of IOL lens
Time Frame: Immediately prior to IOL insertion step of cataract surgery
Population: as for outcome 1
Measure: Number; unit: mm
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 1 | 0
mm |  | 8 |

4. Secondary Outcome: Pupil Size Upon Completion of Surgery
Time Frame: intraoperative
Population: as for outcome 1
Measure: Number; unit: mm
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 1 | 0
mm |  | 7 |

5. Secondary Outcome: Pupil Size on Post-operative Day 1
Time Frame: Post-operative Day 1
Population: Data not available because it wasn't collected
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Patients in Each Arm That Required Another Mydriatic Agent
Time Frame: intraoperative
Population: Data was only collected for the "Intracameral Mydriasis' arm
Measure: Number; unit: percent of participants
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 2 | 0
percent of participants |  | 0 |

7. Secondary Outcome: Cumulative Energy Dispersed for Each Arm
Description: The amount of energy needed to break up the cataractous lens
Time Frame: During cataract surgery
Population: as for outcome 1
Measure: Number; unit: Percent-seconds
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 1 | 0
Percent-seconds |  | 6.6 |

8. Secondary Outcome: Mean Time Taken to Perform Phacoemulsification in Each Arm
Time Frame: intraoperative
Population: as for outcome 1
Measure: Number; unit: seconds
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 1 | 0
seconds |  | 76 |

9. Secondary Outcome: Percentage of Patients With an Increase in the Blood Pressure or Heart Rate
Time Frame: Baseline
Population: Data not available because data was not collected
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Percentage of Patients With an Increase in the Blood Pressure or Heart Rate
Time Frame: intraoperative
Population: Data not available because data was not collected
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Mean Time Taken to Perform Phacoemulsification
Time Frame: During cataract surgery
Population: Data was only collected for the "Intracameral Mydriasis' arm We analyzed data for 1 participant only because of lack of data for the other participant.
Measure: Number; unit: seconds
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 1 | 0
seconds |  | 76 |

12. Secondary Outcome: Percentage of Patients in Each Arm That Required Use of an Iris Expansion Device During the Procedure
Time Frame: intraoperative
Population: Data was only collected for the "Intracameral Mydriasis' arm
Measure: Number; unit: percent
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
Number analyzed (Participants) | 0 | 2 | 0
percent |  | 50 |

ADVERSE EVENTS:
Time Frame: 3 months
Description: Patients not enrolled
Arm/Group | Topical Mydriasis | Intracameral Mydriasis | Topical + Intracameral Mydriasis
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT02909140/Prot_SAP_000.pdf